CLINICAL TRIAL: NCT03300518
Title: A Randomized Study to Analysis the Effectiveness of Estradiol Valerate Pretreatment in Antagonist Protocol for Poor Ovarian Response Patient
Brief Title: Effectiveness of Estradiol Valerate Pretreatment in Antagonist Protocol for Poor Ovarian Response Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSD-MISP-ZX-01
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility
Keywords: GnRH antagonist; Estrogen pretreatment; Poor response patient
MeSH Terms: conditions — Infertility | interventions — follitropin beta; ganirelix; Ovidrel; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pretreatment group (Other): the pretreatment group underwent a modified treatment protocol with pretreatment with estogen administering during the cycle preceding the IVF/ICSI cycle. daily dose of 4 mg (2 mg twice a day) estradiol valerate was given orally in the middle luteal phase which is confirmed seven days after ovulation monitoring by the ultrasound up to 2 days of the next menstrual cycle.Recombinant FSH (Puregon) was initiated on menstrual cycle day 2- 3 at an initial dose of 300 IU/day.A daily administration of ganirelix (0.25 mg Orgalutran; Organon) was introduced when the leading follicle is near 13mm, and was repeated up to the time of hCG administration.Ovulation was triggered when the leading follicles reach 18-20mm and at least two follicles 17-18mm , HCG 10000 IU is used to trigger.
  Interventions: Drug: Follitropin Beta;MSD; Drug: Ganirelix; Drug: hCG; Drug: estradiol valerate
- control groups (Other): In the control groups standard GnRH-antagonist protocol was applied.Recombinant FSH (Puregon) was initiated on menstrual cycle day 2- 3 at an initial dose of 300 IU/day.A daily administration of ganirelix (0.25 mg Orgalutran; Organon) was introduced when the leading follicle is near 13mm, and was repeated up to the time of hCG administration.Ovulation was triggered when the leading follicles reach 18-20mm and at least two follicles 17-18mm , HCG 10000 IU is used to trigger.
  Interventions: Drug: Follitropin Beta;MSD; Drug: Ganirelix; Drug: hCG

INTERVENTIONS:
Drug: Follitropin Beta;MSD — Patients will start stimulation with a daily s.c. injection of follitropin beta( 300IU Puregonon;MSD) menstrual cycle day 2 or 3.
  Other Names: Puregon
Drug: Ganirelix — A daily administration of ganirelix (0.25 mg Orgalutran; MSD) was introduced when the leading follicle is near 13mm, and was repeated up to the time of hCG administration.
  Other Names: Orgalutran
Drug: hCG — Ovulation was triggered when the leading follicles reach 18-20mm and at least two follicles 17-18mm , HCG 10000 IU is used to trigger
  Other Names: Ovidrel
Drug: estradiol valerate — Estradiol valerate (progynova,Schering) daily dose of 4 mg (2 mg twice a day) was given orally, started 7 days before the presumed onset of menses and administered up to 2 days of the next menstrual cycle
  Other Names: progynova
  Arms: pretreatment group

SUMMARY:
The purpose of study is to assess the efficacy of add-on estrogen pretreatment in GnRH antagonist protocol on oocyte retrieval as compared with GnRH antagonist protocol for patients with poor ovarian response Add-on estrogen pretreatment protocol is superior to none pretreatment GnRH antagonist protocol for the number of oocytes retrieval

DETAILED DESCRIPTION:
Women of advanced maternal age seeking ART treatment are characterized as poor ovarian responders in the process of ovarian simulation. Poor response to ovarian stimulation causes high cycle cancellation rate and extremely low pregnancy rate.

More attention has been paid to the potential interest of steroid pretreatments in GnRH antagonist cycles; not only for scheduling the GnRH antagonist cycles, but also for synchronizing the follicular growth which may result in more oocytes retrieved. But available clinical results are controversial.

Previous studies have shown that utilizing the natural negative feedback of the hypothalamus-pituitary-ovary axis induced by estradiol valerate pretreatment effectively prevented inter-cycle increases in follicle-stimulating hormone, improved follicle synchronization, and resulted in a more coordinated follicular development, leading to the recovery of more mature oocytes. However none of the randomized controlled studies compared estradiol valerate pretreatment or not on treatment outcomes, ongoing pregnancy rate, directly on poor response patients using estradiol valerate pretreatment in GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:Bologna criteria

* At least two of the following three features must be present:

  1. Advanced maternal age (≥40 years) or any other risk factor for POR
  2. A previous POR (≤3 oocytes with a conventional stimulation protocol)
  3. An abnormal ovarian reserve test (i.e. antral follicle count < 5-7 follicles or AMH< 0.5 - 1.1 ng/mL)

Exclusion Criteria:

1. Age ≥45 years,
2. Patients who conducted PGD/PGS, and donor egg cycles were excluded.
3. Presence of unilateral ovary absence
4. Abnormal uterine deformity or structure.
5. Spontaneous abortion patients with three or more (including biochemical pregnancy abortion)
6. With other endocrine disease, ovulation disorders such as adrenal cortex function or thyroid dysfunction
7. Have assisted reproductive technology contraindications or pregnancy contraindication of patients

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 552 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
The number of oocytes retrieved by the IVG 36 hours after hCG administration | 36 hours after hCG administration
  The total MII oocytes retrievedd

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6weeks
  clinical pregnancy, defined as intrauterine pregnancy with a positive heartbeat at 6 weeks of gestation.Clinical pregnancy rate:Number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles, or embryo transfer cycles. When clinical pregnancy rates are given, the denominator must be specified.
ongoing pregnancy rate | 12weeks
  ongoing pregnancy defined as an intact pregnancy at 12 weeks of gestation
Optimal number of embryo | 1 week
  According to the embryonic developmental rate and morphology, the high quality embryos were defined as the next day (D2) transplanted embryos reached 3 or 4 cells and the third day (D3) transplanted embryos reached 6 to 8 cells with morphological grade 1 or 2

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gong, Doctor, Study Director — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of Citic-Xiangya, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang S, Tang Y, Wang X, Zong Y, Li X, Cai S, Ma H, Guo H, Song J, Lin G, Lu G, Gong F. Estrogen valerate pretreatment with the antagonist protocol does not increase oocyte retrieval in patients with low ovarian response: a randomized controlled trial. Hum Reprod. 2022 Jun 30;37(7):1431-1439. doi: 10.1093/humrep/deac081. PMID 35460400